CLINICAL TRIAL: NCT06673394
Title: Eculizumab For Acute Attack of Neuromyelitis Optica Spectrum Disorder (NMOSD): a Multi-Center, Phase 2, Open Label Trial (EASE-NMO)
Brief Title: Eculizumab For Acute Attack of Neuromyelitis Optica Spectrum Disorder
Acronym: EASE-NMO
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study plan need to be modified after widely discussion with our consultation board, regarding the conscern about the efficiency may not be able to detect the expected differences. We would like to withdraw this study plan and startup a new one.
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Fu-Dong Shi, Professor, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EASE-NMO
Record Dates: First submitted 2024-10-30; First posted 2024-11-04 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2024-11

CONDITIONS: Neuromyelitis Optica Spectrum Disorder Attack
Keywords: Eculizumab; Acute Attack; Neuromyelitis Optica Spectrum Disorder
MeSH Terms: conditions — Neuromyelitis Optica | interventions — eculizumab; Methylprednisolone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IVMP arm (Other): IVMP arm: 1000mg methylprednisolone x5d, oral prednisone 60mg, 5mg weekly decline + antibiotics
  Interventions: Drug: IVMP
- eculizumab arm (Active Comparator): Eculizumab arm: eculizumab (900 mg) will be administered intravenously once per week for a total of four doses (days 1, 8, 15, and 22) in conjunction with IVMP and oral prednisone (60mg, 5mg weekly decline). Terminal complement complex inhibition by eculizumab predisposes patients to infections by encapsulated bacteria, especially N meningitidis. Meningococcal vaccination will not be effective in this timeframe; instead, all enrolled patients will receive antibiotic prophylaxis against N meningitidis from the time of the first dose of the study drug to 8 weeks after the last administration
  Interventions: Drug: Complement protein C5 inhibitor; Drug: IVMP

INTERVENTIONS:
Drug: Complement protein C5 inhibitor — Investigational arm: eculizumab (900 mg) will be administered intravenously once per week for a total of four doses (days 1, 8, 15, and 22) in conjunction with IVMP and oral prednisone (60mg, 5mg weekly decline). Terminal complement complex inhibition by eculizumab predisposes patients to infections by encapsulated bacteria, especially N meningitidis. Meningococcal vaccination will not be effective in this timeframe; instead, all enrolled patients will receive antibiotic prophylaxis against N meningitidis from the time of the first dose of the study drug to 8 weeks after the last administration.
  Other Names: eculizumab
  Arms: eculizumab arm
Drug: IVMP — IVMP arm: 1000mg methylprednisolone x5d, oral prednisone 60mg, 5mg weekly decline + antibiotics
  Other Names: methylprednisolone; prednisolone

SUMMARY:
Neuromyelitis optica spectrum disorder (NMOSD) is a relapsing, inflammatory autoimmune disorder of the central nervous system characterized by the pathogenic anti-aquaporin 4 antibody (AQP4-IgG). The objectives of this study are to assess the efficacy and safety of eculizumab for treatment of patients with neuromyelitis optica spectrum disorders during acute phase who are anti-aquaporin-4 (AQP4) antibody-positive. Eculizumab, a humanized monoclonal antibody, inhibits the terminal complement protein C5 and prevents its cleavage into C5a and the formation of C5b-9 (MAC), has approved for preventive treatment of NMOSD. Given the high efficacy of C5 inhibition, eculizumab is proposed to potentially provide rapid relief from astrocyte destruction by reducing MAC formation, which could contribute to the fast alleviation of neurological deficit during NMO acute attack. The potential of eculizumab warrants further investigation as a treatment for acute neuromyelitis optica spectrum disorders attacks.

ELIGIBILITY:
Inclusion criteria:

1. Anti-AQP4 antibody seropositive.
2. Male or female patients ≥18 years old
3. Body weight ≥ 35 kg
4. Leukocyte and CRP in the normal range
5. Acute optic neuritis and/or transverse myelitis presenting to the hospital within 10 days of symptom onset. An acute CNS inflammatory attack is defined as:

   • An acute presentation of neurological symptoms evolving over the course of 4 hours to 21 days that i. Localize to the spinal cord such as weakness, numbness or bowel/bladder dysfunction; or ii. Localize to the optic nerve with loss of visual acuity

   • Associated with a change in neurological exam that meet the following thresholds: i. Spinal cord lesions must show a reduction in 1 point on the EDSS scale from baseline; or a reduction of 0.5 if baseline EDSS is at least 5.5.

   ii. Optic nerve lesions must show a reduction in visual acuity by at least 2 lines on the vision chart.

   • Also associated with any of the following objective findings: i. New gadolinium-enhancing MRI lesion in the area of the CNS that correlates with the exam findings, or ii. Cerebrospinal fluid findings of pleocytosis with at least 10 WBC per microliter, or iii. Swelling of the optic nerve head on fundoscopy or swelling of the retinal nerve fiber layer by OCT of at least 25 microns from baseline.
6. A female subject is eligible to enter the trial if she is:

   * Not pregnant or nursing;
   * Of non-childbearing potential (i.e. women who have had a hysterectomy, are post-menopausal, which is defined as >2 years without menses or, in female subjects who have been post-menopausal for <2 years, must be confirmed with Follicle Stimulating Hormone (FSH) and estradiol levels), have both ovaries surgically removed or have current documented tubal ligation) OR
   * Of child-bearing potential (i.e. women with functional ovaries and no documented impairment of oviductal or uterine function that would cause sterility). This category includes women with oligomenorrhoea (even severe), women who are perimenopausal or have just begun to menstruate.
   * Subject has a negative serum pregnancy test at screening and agrees to one of the following:

     i. Complete abstinence from intercourse for the period from consent to trial until 6. months after the last dose of investigational product; or, ii. Consistent and correct use of one of the following acceptable methods of birth control for the period from consent into the trial until 6 months after the last dose of investigational product: i.Oral contraceptives (either combined or progesterone only) ii. Injectable progesterone iii. Levonorgestrel implants iv. Estrogenic vaginal ring v. Percutaneous contraceptive patches vi.Intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of <1% per year vii.Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the trial; this male must be the sole partner for the subject viii.Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository).

Exclusion criteria:

1. Current evidence or known history of clinically significant infection including:

   * Chronic or ongoing active infectious disease requiring long term systemic treatment such as, but not limited to: PML, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis, or active hepatitis C
   * Previous serious opportunistic or atypical infections
   * History of positive serology for hepatitis B (unless history of vaccination)
   * Prior history, or suspicion, of tuberculosis (TB)
   * History of positive serology for HIV
   * Past or current history of medically significant adverse effects (including allergic reactions) from: Corticosteroids / Eculizumab
2. Current malignancy or history of malignancy in remission within the past 5 years, except for

   * Cervical carcinoma Stage 1B or less
   * Non-invasive basal cell and squamous cell skin carcinoma
   * Cancer diagnoses with a duration of complete response (remission) >5 years
3. Significant concurrent, uncontrolled medical condition including, but not limited to, cardiac, renal, hepatic, hematological, gastrointestinal, endocrine, immunodeficiency syndrome, pulmonary, cerebral, psychiatric, or neurological disease which could affect the subject's safety, impair the subject's reliable participation in the trial, impair the evaluation of endpoints, or necessitate the use of medication not allowed by the protocol, as determined by the principal investigator of the trial.
4. Use of an investigational drug or other experimental therapy within 4 weeks, 5 pharmacokinetic half-lives or duration of biological effect (whichever is longer) prior to screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09-03 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Mean change in OSIS from presentation to Day 28 | Acute attack to week4
  The Optic-Spinal Impairment Score (OSIS) was developed to measure the disability status of subjects with demyelinating disease. It allows an objective quantification of the level of functioning that could be widely and reproducibly used by researchers and health care providers. The OSIS evaluates four primary functions: Visual Acuity (VA) (0-8), Motor Function (0-7), Sensory Function (0-5), and Sphincter Function (0-5). A higher OSIS score indicates a more severe level of disability. The standards for the OSIS scoring are as follows:
  Optic-Spinal Impairment Score (OSIS) Visual Acuity (VA) 0 Normal
  1. Scotoma but VA (corrected) better than 20/30
  2. VA 20/30-20/59
  3. VA 20/60-20/100
  4. VA 20/I0I-2012004
  5. VA 20/20I-20/800.
  6. Count fingers only
  7. Light perception only
  8. No light perception Motor Function
  0 Normal
  1. Abnormal signs (hyperreflexia, Babinski sign) without weakness
  2. Mild weakness (MRC grade 5-or 4+) in affected limb(s)
  3. Mo

SECONDARY OUTCOMES:
Change in EDSS from presentation to Day 28 | Acute attack to week4
  The Kurtzke Expanded Disability Status Scale (EDSS) was developed to measure the disability status of subjects with demyelinating disease. It allows an objective quantification of the level of functioning that could be widely and reproducibly used by researchers and health care providers. The EDSS provides a total score on a scale that ranges from 0 to 10 where 0 is normal and 10 is deceased. Increasing disability is reflected in an increasing EDSS score.

IPD SHARING:
Plan to Share IPD: No